CLINICAL TRIAL: NCT06542640
Title: Identifying Mechanisms of Response to Therapeutic Intervention in Clinical High Risk (CHR) for Psychosis: a Bridge to Treatment
Brief Title: Mechanisms of Response to Therapeutic Intervention in Clinical High Risk (CHR) for Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Florida A&M University (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); VA Boston Healthcare System (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, William Stone, Associate Professor of Psychology in the Department of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2023P001089; 2R01MH111448 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-08-07 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Psychosis; Schizophrenia-Like; Healthy Controls
Keywords: real-time fMRI neurofeedback (rt-fMRI-NFB); mindfulness-based (mb); mb rt-fMRI-NFB (mb-rt-fMRI-NFB); repet. transcran mag stim (rTMS); neuropsycho (NP); diffusion tensor imaging (DTI); clinical high risk (CHR); healthy control (HC); MATRICS Consenus Cog Batt (MCCB)
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The study will consist of two interventions and 2 full assessments, (pre- and post-intervention) (year 1) followed by two clinical/NP/NLP/ERP assessments in years 2 and 3 relative to a CHR's entry to the study. To minimize the time lag between HC's assessment and the last follow-up assessment of the CHR, 50 HC participants will be recruited at the study onset and 50 additional HC will be recruited at years 3 and 4 of the grant. Baseline assessments will be followed by random assignment of CHR subjects to either an intervention group (100 CHR) or sham group (100 CHR). The intervention group will receive either the TMS (50 CHR) or rt-fMRI NFB (50 CHR), with the random CHR assignment to the arm of the study. The sham groups will also be counterbalanced across subjects, with 50 CHR in the TMS-sham and 50 CHR in the rt-fMRI NFB-first group. The two interventions will be delivered over two-week period, followed by post-intervention assessments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and investigators will be blinded to whether participants at CHR for psychosis are randomized to either the real treatment or to the sham conditions for either of the mb-rt-fMRI-NFB or the rTMS conditions. Similarly, outcomes assessors and clinical care providers will be blinded as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CHR with mb-rt-fMRI-NFB Group (Experimental): This CHR group will receive experimental treatment via mb-rt-fMRI-NFB, in a targeted frontal lobe region including the dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Mb-rt-fMRI-NFB
- CHR with sham mb-rt-fMRI-NFB Group (Sham Comparator): This CHR group will receive treatment via mb-rt-fMRI-NFB, but in a different, uninvolved brain region
  Interventions: Device: Sham mb-rt-fMRI-NFB
- CHR with rTMS Group (Experimental): This CHR group will receive experimental treatment via rTMS, along a targeted neural pathway extending from the cerebellum to the midbrain to the dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: rTMS
- CHR with sham rTMS Group (Sham Comparator): This CHR group will receive treatment via rTMS, but in a different, uninvolved brain region
  Interventions: Device: Sham rTMS
- Healthy Control Group (No Intervention): The healthy control group will not receive any treatment, but will be used as a comparison for the 2 experimental and 2 sham groups.

INTERVENTIONS:
Device: Mb-rt-fMRI-NFB — The MRI and TMS interventions described below will yield measures of change in the targeted brain regions in post- relative to pre- intervention comparisons. These change measures will be compared relative to changes in the sham/control group and the HC group. Furthermore, they will be compared to HC to assess improvement or normalization of brain function in the targeted brain regions. In addition, the investigators will examine treatment effects on traditional biomarkers that are likely to be impacted by such interventions: ERP, NP and NLP measures. Here, mindfulness meditation practiced during a real-time fMRI NFB session will be used to bring connectivity changes to brain structures involved in positive psychiatric symptoms (e.g. attenuated psychotic symptoms) in order to to reduce them.
  Arms: CHR with mb-rt-fMRI-NFB Group
Device: Sham mb-rt-fMRI-NFB — Individuals with CHR who are randomly assigned to this arm will receive mb-rt-fMRI-NFB, as do the experimental group, but it will be aimed at a motor cortex location that is not part of the prefrontal neural networks targeted in the experimental group.
  Arms: CHR with sham mb-rt-fMRI-NFB Group
Device: rTMS — In previous work, the investigators used a multivariate pattern analysis to identify functional connectivity correlates of negative symptom severity in a schizophrenia (SZ) group. DLPFC-cerebellum hypo-connectivity was strongly correlated with negative symptoms. In a separate SZ cohort, the investigators used rTMS targeting the cerebellum to manipulate this circuit. The rTMS-induced increase in functional connectivity in a cerebellar-midbrain-DLPFC circuit was strongly linked to negative symptom severity reduction. Furthermore, individuals varied in the degree of change in functional connectivity in response to rTMS. This variation strongly predicted variation in post-rTMS symptom severity. The investigators predict that rTMS based intervention, but not sham rTMS, will similarly impact the cerebellar-midbrain-dorsolateral prefrontal cortex (DLPFC) network in the CHR group receiving real but not sham rTMS.
  Arms: CHR with rTMS Group
Device: Sham rTMS — Individuals with CHR who are randomly assigned to this arm will receive rTMS, as do the experimental group, but it will be aimed at a motor cortex location that is not part of the prefrontal neural networks targeted in the experimental group.
  Arms: CHR with sham rTMS Group

SUMMARY:
This study, "Psychobiological Follow-up Study of Transition from Prodrome to Early Psychosis", will be conducted in collaboration with the Shanghai Mental Health Center (SMHC) and several data processing sites in the United States. The current study builds on findings from the investigator's previous work that identified several biomarkers in participants at clinical high risk (CHR) for psychosis that may be related to clinical outcomes such as the development of psychosis. This study responds to the critical need to understand links between biomarkers (could be clinical, cognitive, biological or other abnormalities) and later clinical outcomes.

Participants will receive either one of two real interventions or one of two sham (a procedure that looks like the real treatment but is not) interventions, involving either: 1. repetitive transcranial magnetic stimulation (rTMS)1; or 2. mindfulness-based real time fMRI neurofeedback (mb-rt-fMRI-NFB). Both procedures will measure brain capacity for change in CHR individuals, thus paving the way forward for future therapeutic interventions.

The main hypotheses to be addressed by this study are:

1. - Following real interventions, novel biomarkers will be more effective predictors of clinical outcome than standard biomarkers in participants at CHR for psychosis
2. - Following real interventions, novel biomarkers will be more effective predictors of clinical outcomes in participants who received the real intervention than in participants who received sham treatments
3. - The novel interventions will reduce biomarker abnormalities in individuals with CHR relative to their own baselines and relative to healthy controls (HC)
4. - The sham interventions will will not reduce biomarker abnormalities in individuals with CHR relative to their own baselines or relative to HC

DETAILED DESCRIPTION:
This study builds upon our previous work, entitled "Psychobiological Follow-up Study of Transition from Prodrome to Early Psychosis" (R01MH111448). This study, titled Mechanisms of Response to Therapeutic Intervention in Clinical High Risk (CHR) for Psychosis: A bridge to treatment", focuses on two persistent needs in clinical high risk (CHR) for psychosis research: 1) the identification of novel biomarkers associated with transition to psychosis and other clinical outcomes; and 2) the identification of symptom-specific brain circuit targets that can be engaged in future clinical trials. The investigators hypothesize that clinically relevant biomarkers for participant-specific prognosis in CHR will be enhanced by the inclusion of biomarker measures that allow for the quantitative assessment of neural plasticity and are likely amenable to therapeutic change. In this view, CHR clinical outcomes are likely determined by both pathophysiology and by the brain's capacity to adapt and respond to pathophysiology via neural plasticity mechanisms. The investigators thus propose to examine brain circuit plasticity biomarkers relevant to CHR by administering non-invasive neuromodulation via two novel paradigms that, as they demonstrated previously in schizophrenia, engage brain networks involved in negative and positive psychiatric symptoms. These two novel interventional techniques are: 1. repetitive transcranial magnetic stimulation (rTMS); and 2. mindfulness-based real time functional magnetic resonance imaging (rt-fMRI) neurofeedback enhanced mindful meditation (mb-rt-fMRI-NFB) The investigators will also collect both traditional biomarkers (for example, clinical, neuropsychological, electrophysiological and neuroimaging biomarkers) and the novel biomarkers listed above (i.e., biomarkers that quantify neural changes pre- relative to post-intervention). These two interventions, which have not been used with CHR subjects before, will be tested in 200 CHR (50 CHR per experimental condition) and 100 HC over 5 years. Furthermore, the investigators will continue to enhance knowledge capacity at the Shanghai Mental Health Center (SMHC), where their Chinese collaborators are based. They will also examine the effectiveness of these interventions in CHR as a bridge to future therapeutic treatments and will test traditional and novel biomarkers as predictors of clinical and neurocognitive outcomes. Additionally, the investigators will significantly enhance research capacity by building on already established achievements and collaborations, and by extending their reach to new institutions (Aim 4). This competitive renewal capitalizes on a unique set of strengths at a single site (SMHC) and on a collaboration with the Shanghai research team, which has proven to be most productive in the current grant cycle. The investigators hypothesize that this highly novel study will contribute to the development of future therapeutic interventions in CHR, which will prevent this vulnerable population from developing adverse outcomes and, at the same time, will enrich the CHR field with new insights into the pathophysiology of this condition.

ELIGIBILITY:
Inclusion Criteria:

Clinical High Risk (CHR):

1. Male or female between 15 and 35 years old.
2. Can understand and sign an informed consent (or assent for minors) document.
3. Must meet the substance use criteria:

   1. No Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) Alcohol or Drug Dependence in the past 3 months;
   2. No use on the day of assessment, clearly not intoxicated or hung-over.
4. Must meet diagnostic criteria for a prodromal syndrome. If under the age of 19 and meet diagnostic criteria for Schizotypal Personality Disorder or meet the diagnostic criteria called the Criteria for Prodromal Syndromes (COPS), which are operationalized as follows (a-c below):

   1. Genetic Risk and Deterioration Syndrome (GRDS): First degree biological relative with psychosis or subject with Schizotypal Personality Disorder and a 30% drop in Global Assessment of Functioning (GAF) score compared to one year ago, sustained over the past month.
   2. Attenuated Positive Symptoms Syndrome (APSS): Severity rating of moderate (rating of 3), moderately severe (4) or severe but not psychotic (5) on any one of the five Symptoms of Psychotic Disorders (SOPS) positive symptoms; symptom occurs at or above moderate severity level at an average frequency of at least once per week in the past month; symptom must have begun in the past year or currently rates at least one scale point higher than rated 12 months previously.
   3. Brief Intermittent Psychotic Syndrome (BIPS): Severity rating of psychotic intensity (6) on any of the 5 SOPS positive symptoms; symptom is present at least several minutes per day at a frequency of at least once per month; symptom(s) must have reached a psychotic intensity in the past 3 months; symptom is not seriously disorganizing or dangerous; symptom(s) do not last for more than 1 hour/day at an average frequency of 4 days/week over 1 month.
5. . Participant may be remitted from the CHR syndrome or may have converted to a full psychotic disorder since study entry and either is acceptable - they remain eligible to participate in follow-up procedures.

Exclusion Criteria:

1. Meet criteria for current or lifetime Axis I psychotic disorder, including affective psychoses and psychosis Not Otherwise Specified (NOS) at the baseline assessment
2. Impaired intellectual functioning (i.e., Intelligence Quotient (IQ)<70) at baseline.
3. Past history of or current clinically significant central nervous system disorder that may contribute to prodromal symptoms or confound their assessment.
4. Traumatic Brain Injury that is rated as 7 or above on the Traumatic Brain Injury screening instrument (signifying a significant brain injury with persistent sequelae) or current concussion that interferes with any assessment measures.
5. Diagnostic prodromal symptoms that are clearly caused by one or more other psychiatric disorders, including substance use disorders, in the judgment of the evaluating clinician. Other non-psychotic Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) disorders will not be exclusionary (e.g., substance abuse disorder, major depression, anxiety disorders, personality disorders), as long as the disorder does not account for the diagnosis of prodromal symptoms.

Healthy Controls (HC):

1. Must meet subject inclusion criteria 1-2 and exclusion criteria 1-5. Must not meet criteria for any prodromal syndrome, any current or past psychotic disorder or Cluster A personality disorder diagnosis and must not be receiving any current treatment with psychotropic medication at the baseline assessment.
2. Must not have a family history (in first-degree relatives) of schizophrenia, schizoaffective disorder, schizotypal personality disorder, or any other disorder involving psychotic symptoms.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
mb-rt-fMRI-NFB intervention: functional connectivity | 1 month, 1 year, 2 years
  Context-dependent changes in functional connectivity (i.e., coupling) between brain regions will be measured by statistical software programs as Pearson correlation coefficients between brain regions whose activity depends on an interaction between psychological context (the task) and physiological state (the time course of brain activity)
rTMS intervention: functional connectivity | 1 month, 1 year, 2 years
  Context-dependent changes in functional connectivity (i.e., coupling) between brain regions will be measured by statistical software programs as Pearson correlation coefficients between brain regions whose activity depends on an interaction between psychological context (the task) and physiological state (the time course of brain activity)

SECONDARY OUTCOMES:
Clinical | 1 month, 1 year, 2 years
  Changes in Clinical High Risk clinical function from baseline will measured using the Structured Interview for Psychosis Risk Syndromes, specifically the Scale for Psychosis Risk Symptoms and the Criteria for Psychosis Risk Syndromes
Neuropsychological function: verbal learning | 1 month, 1 year, 2 years
  Changes in verbal learning from baseline will be measured in the Clinical High Risk participants using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery: Hopkins Verbal Learning Test - Revised
Neuropsychological function: visual learning | 1 month, 1 year, 2 years
  Changes in visual learning from baseline will be measured in the Clinical High Risk participants using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery: Brief Visuospatial Memory Test - Revised
Neuropsychological function: visual-spatial / speed of processing | 1 month, 1 year, 2 years
  Changes in visual-spatial speed of processing from baseline will be measured in the Clinical High Risk participants using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery: Trail Making Test
Neuropsychological function: verbal fluency / speed of processing | 1 month, 1 year, 2 years
  Changes in verbal fluency / speed of processing from baseline will be measured in the Clinical High Risk participants using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery: Category Fluency: Animal Naming Test
Neuropsychological function: visual-motor / speed of processing | 1 month, 1 year, 2 years
  Changes in visual-motor / speed of processing from baseline will be measured in the Clinical High Risk participants using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery: Brief Assessment of Cognition in Schizophrenia: Symbol Coding
Neuropsychological function: attention | 1 month, 1 year, 2 years
  Changes in attention from baseline will be measured in the Clinical High Risk participants using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery: Continuous Performance Test: Identical Pairs Version
Neuropsychological function: working memory | 1 month, 1 year, 2 years
  Changes in working memory from baseline will be measured in the Clinical High Risk participants using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery: Wechsler Memory Scale - Third Edition: Spatial Span
Neuropsychological function: reasoning and problem solving | 1 month, 1 year, 2 years
  Changes in reasoning and problem solving from baseline will be measured in the Clinical High Risk participants using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery: Neuropsychological Assessment Battery: Mazes
Event Related Potentials | 1 month, 1 year, 2 years
  Changes in Clinical High Risk participant's electrophysiological function from baseline will be measured through measures of wave amplitudes and latencies in 'P300 Oddball' and 'P300 Novel' paradigms
Natural Language Processing: Linguistic | 1 month, 1 year, 2 years
  Changes in Clinical High Risk participant's natural language function from baseline will be measured linguistically using machine learning: semantic coherence
Natural Language Processing: Acoustic | 1 month, 1 year, 2 years
  Changes in Clinical High Risk participant's natural language function from baseline will be measured acoustically using machine learning: pauses in words
Structural MRI | 1 month, 1 year, 2 years
  Changes in Clinical High Risk participant's cortical gray matter brain function will be measured through cortical thickness
Diffusion Tensor Imaging | 1 month, 1 year, 2 years
  Changes in Clinical High Risk participant's brain white matter function will be measured using 'fractional anisotropy', which is a measurement of the directionality of water diffusion in white matter, which is used in diffusion imaging to assess the density of white matter fibers, axonal diameter, and myelination

CONTACTS AND LOCATIONS:
Overall Officials: William S Stone, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data, which will not contain Protected Health Information (PHI), will be transmitted from the Shanghai site to the U.S. sites. All human-subjects data provided will include a Global Unique Identifier (GUID) and will not include personally identifiable information (PII). Descriptive/raw data are data used to characterize a research subject, will include data from standard diagnostic assessments, standard clinical measures, demographic data, and will be submitted to New Drug and Clinical Trials rules (NDCT). Analyzed data will be submitted prior to publication/public dissemination (whether the findings are positive or negative). Even if a publication focuses on only part of an analyzed dataset, the entire analyzed dataset will be submitted when the first paper/finding is published or communicated. The data that are not part of the paper will not be immediately shared, but rather along the time frame described below.
Time Frame: Data will be submitted to NDCT on a semi-annual basis (on or before January 15 and July 15, beginning six months after the award budget period has begun). Raw neuroimaging data will be submitted incrementally as new data are acquired. Descriptive/raw research data are held until the finding is communicated or published. Analyzed data are expected at the time a manuscript is accepted for publication. These data will then be shared when the publication is released, along with the associated descriptive data. Data that remain unpublished are expected prior to project completion and will be shared within one year after the original project completion date, allowing the Principal Investigator and his/her team sufficient time to complete appropriate quality assurance/quality control procedures.
Access Criteria: All submitted data (both descriptive/raw and analyzed data) will be made available for access by qualified members of the research community according to the provisions defined in the National Institute of Mental Health (NIMH) Data Repositories Data Access Agreement and Use Certification. These procedures are intended to allow investigators sufficient time for data verification, and for submission of primary publications based on the collected data.

REFERENCES:
- [Background] Brady RO Jr, Gonsalvez I, Lee I, Ongur D, Seidman LJ, Schmahmann JD, Eack SM, Keshavan MS, Pascual-Leone A, Halko MA. Cerebellar-Prefrontal Network Connectivity and Negative Symptoms in Schizophrenia. Am J Psychiatry. 2019 Jul 1;176(7):512-520. doi: 10.1176/appi.ajp.2018.18040429. Epub 2019 Jan 30. PMID 30696271
- [Background] Okano K, Bauer CCC, Ghosh SS, Lee YJ, Melero H, de Los Angeles C, Nestor PG, Del Re EC, Northoff G, Whitfield-Gabrieli S, Niznikiewicz MA. Real-time fMRI feedback impacts brain activation, results in auditory hallucinations reduction: Part 1: Superior temporal gyrus -Preliminary evidence. Psychiatry Res. 2020 Apr;286:112862. doi: 10.1016/j.psychres.2020.112862. Epub 2020 Feb 10. PMID 32113035
- [Background] Bauer CCC, Okano K, Ghosh SS, Lee YJ, Melero H, Angeles CL, Nestor PG, Del Re EC, Northoff G, Niznikiewicz MA, Whitfield-Gabrieli S. Real-time fMRI neurofeedback reduces auditory hallucinations and modulates resting state connectivity of involved brain regions: Part 2: Default mode network -preliminary evidence. Psychiatry Res. 2020 Feb;284:112770. doi: 10.1016/j.psychres.2020.112770. Epub 2020 Jan 14. PMID 32004893
- [Result] Niznikiewicz MA, Brady RO, Whitfield-Gabrieli S, Keshavan MS, Zhang T, Li H, Pasternak O, Shenton ME, Wang J, Stone WS. Dynamic intervention-based biomarkers may reduce heterogeneity and motivate targeted interventions in clinical high risk for psychosis. Schizophr Res. 2022 Aug;246:60-62. doi: 10.1016/j.schres.2022.05.004. Epub 2022 Jun 13. No abstract available. PMID 35709648